CLINICAL TRIAL: NCT04686253
Title: Internal Microstructure of Patent Foramen Ovale Related to Cryptogenic Stroke, Transient Ischemic Attack or Migraine
Brief Title: Internal Microstructure of Patent Foramen Ovale Related to Stroke
Acronym: IMPORT
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Beijing Anzhen Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Tibet Autonomous Region People's Hospital (Other); Beijing Tiantan Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-6
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Patent Foramen Ovale
Keywords: patent foramen ovale; stroke; transient ischemic attack; migraine; microstructure
MeSH Terms: conditions — Foramen Ovale, Patent; Stroke; Ischemic Attack, Transient; Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PFO patients with CS or/and TIA: PFO patients with CS or/and TIA (transcatheter closure of PFO was performed).
  Interventions: Other: not appliable
- PFO patients with migraine: PFO patients with migraine (transcatheter closure of PFO was performed).
  Interventions: Other: not appliable
- PFO patients without symptom: PFO patients without symptom (5-year follow-up).
  Interventions: Other: not appliable

INTERVENTIONS:
Other: not appliable — not appliable

SUMMARY:
This study aims to (1) investigate the internal microstructure of patent foramen ovale related to cryptogenic stroke, transient ischemic attack or migraine and determine the effectiveness of transcatheter closure in these patients; (2) evaluate the microstructural features of asymptomatic patients with PFO and make a follow-up；(3) perform an untargeted metabolomics analysis using plasma samples from right atrium and left atrium and shunt provocative test was conducted;(4) collect the blood sample from PFO tunnel;(5) cardiac CTA was performed to evaluate the position and morphology of device.

DETAILED DESCRIPTION:
Patent foramen ovale (PFO) is associated with a variety of pathological conditions, and it is presumed to be related to the occurrence of cryptogenic stroke (CS), transient ischemic attack (TIA) or migraine. In addition, the main hypothesized pathophysiologic mechanism is paradoxical embolization, namely microemboli or metabolites from the venous circulation to enter the systemic circulation. The morphological characteristics of PFO have the potential to predict risks and screen the appropriate candidates for transcatheter closure. The structure features for predicting risk included atrial septal aneurysm, a large right-left shunt, long-tunnel PFO and so on. However, the in-vivo internal microstructure of PFO is still unclear. The microstructural features might provide important information for better understanding the PFO and risk stratification.

The aim of this study is to (1) investigate the internal microstructure of patent foramen ovale related to cryptogenic stroke, transient ischemic attack or migraine and determine the effectiveness of transcatheter closure in these patients; (2) evaluate the microstructural features of asymptomatic patients with PFO and make a follow-up；(3) perform an untargeted metabolomics analysis using plasma samples from right atrium and left atrium and shunt provocative test was conducted;(4) collect the blood sample from PFO tunnel;(5) cardiac CTA was performed to evaluate the position and morphology of device.

This study will enroll subjects with PFO, and enrollment will be divided into three phases.

Phase 1: PFO patients with CS or/and TIA (transcatheter closure of PFO was performed). A minimum of 500 patients is reached.

Phase 2: PFO patients with migraine (transcatheter closure of PFO was performed). A minimum of 500 patients is reached.

Phase 3: PFO patients without symptom (5-year follow-up). A minimum of 200 patients is reached.

In addition, blood samples were obtained, including inferior vena cava, superior vena cava, right atrium, PFO-tunnel, left pulmonary artery, left atrium and left pulmonary vein. Then, another 20 ml blood sample was obtained from right atrium (near PFO) and injected into left atrium immediately. During a ten-minute waiting period, any symptom was recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 16 to 65 years without any known vascular risk factor, including hypertension, hypercholesterolemia, diabetes mellitus, atrial fibrillation, smoking and obesity;
2. Documented PFO with right-to-left shunt ≥ 20 micro-bubbles by c-TCD;
3. Stroke group: history of ischemic stroke (based on brain magnetic resonance imaging) or TIA within 6 months without other identifiable causes (Phase1);
4. Migraine group: history of migraine headaches more than one year without other identifiable causes (Phase2);
5. Control group: incidental finding of PFO without neurological or systemic symptoms (Phase3).

Exclusion Criteria:

1. Any identifiable cause of ischemic stroke/TIA or migraine other than PFO;
2. History of stroke or TIA within the past one month;
3. Presence of cardiac enlargement or dysfunction;
4. Presence of coexisting cardiovascular structural malformations/diseases;
5. Presence of carotid artery lesions or coronary artery disease;
6. Presence of deep vein thrombosis or pulmonary embolism;
7. Presence of implanted cardiac devices;
8. Evidence of hypercoagulable state;
9. Allergic to contrast medium;
10. Echocardiographic evidence of intra-cardiac thrombus, mass, tumor or vegetation;
11. Active endocarditis or other infections.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll subjects with PFO, and enrollment will be divided into three cohorts.
  Cohort 1: PFO patients with CS or/and TIA (transcatheter closure of PFO was performed). A minimum of 100 patients is reached.
  Cohort 2: PFO patients with migraine (transcatheter closure of PFO was performed). A minimum of 100 patients is reached.
  Cohort 3: PFO patients without symptom (5-year follow-up). A minimum of 100 patients is reached.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events after evaluation of PFO internal microstructure | 5 years
  cryptogenic stroke, transient ischemic attack , migraine or systemic embolism

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chaowu Yan, Beijing, Beijing Municipality
  - National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences,Fuwai Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yan C, Li H, Wang C, Yu H, Guo T, Wan L, Yundan P, Wang L, Fang W. Frequency and Size of In Situ Thrombus Within Patent Foramen Ovale. Stroke. 2023 May;54(5):1205-1213. doi: 10.1161/STROKEAHA.122.041524. Epub 2023 Mar 9. PMID 36891906
- [Background] Yan C, Li H. Preliminary Investigation of In situ Thrombus Within Patent Foramen Ovale in Patients With and Without Stroke. JAMA. 2021 May 25;325(20):2116-2118. doi: 10.1001/jama.2021.4359. PMID 34032839